CLINICAL TRIAL: NCT03687697
Title: A Randomized Controlled Trial Comparing Global Medium With G-TL, Cornell Single and Sequential Steps Media by the Time-Lapse System.
Brief Title: Comparison of Global, G-TL, & Cornell Media
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was halted prior to enrollment of first participant due to non funding and recourses.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1707018347
Record Dates: First submitted 2018-07-31; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Infertility
Keywords: IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Global vs. G-TL Media (Experimental): Global medium will be compared with G-TL (Time-Lapse) medium.
  Interventions: Biological: Global vs. G-TL vs Cornell's C3 vs Cornell's C1/C2 media
- Global vs. Cornell's C3 Media (Experimental): Global medium will be compared with Cornell's C3 single step medium.
  Interventions: Biological: Global vs. G-TL vs Cornell's C3 vs Cornell's C1/C2 media
- Global vs. Cornell's sequential Media (Experimental): Global medium will be compared with Cornell's C1/C2 sequential medium.
  Interventions: Biological: Global vs. G-TL vs Cornell's C3 vs Cornell's C1/C2 media

INTERVENTIONS:
Biological: Global vs. G-TL vs Cornell's C3 vs Cornell's C1/C2 media — A comparison between Global, G-TL, Cornell's C3, and Cornell's C1/C2 embryo culture media.

SUMMARY:
This is a prospective, randomized clinical trial to compare the Global commercial single step media to 1) G-TL (Vitrolife), 2) Weill Cornell's single step and sequential steps media, which all support human embryo development in the laboratory using the Vitrolife Time-Lapse system. The main goal of the study is to identify the best culture medium for optimal embryo development.

DETAILED DESCRIPTION:
Culture media are used to culture embryos in order to support their development in the laboratory. New media are being introduced to the market. Clinical studies have shown that the use of the single-step Global medium for culture of human embryos from the zygote stage to the blastocyst stage has resulted in better in-vitro development than a variety of sequential media system.

Global is a FDA approved commercial single-step medium for all embryo culture from Day 0 to the blastocyst stage.

G-TL (Time-Lapse) is a FDA approved commercial single-step medium from Vitrolife. It was developed to be used with time-lapse devices as a continuous embryo culture medium from Day 0 to Day 5/6.

C3 is Cornell's in house made single-step buffered medium for embryo culture from oocyte fertilization to blastocyst stage used as standard of care.

C1/C2 is Cornell's in house made buffered sequential medium otherwise known as multi step medium, use to culture embryos for development. It is formulated to meet the embryos requirements at two specific stages of development but require removal of the dish from the incubator to physically exchange the culture media surrounding the embryos. This medium will be the control.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or younger (maternal)
* 65 years of age or younger (paternal)
* 10 or more oocytes
* Fresh or frozen oocytes (including donor)
* Fresh or frozen (including donor) sperm can be used
* ICSI only
* Frozen embryos from this study can be included in the outcome portion of this study.
* PGD and/or PGS patients included

Exclusion Criteria:

* Patients with less than 10 oocytes
* Co-culture patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Maternal age- 40 years of age or younger Paternal age- 65 years of age or younger
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Embryo development | Day 5
  Comparison of embryo development using standard assessments of morphology, cell number, and embryo grading, between the different media groups.

SECONDARY OUTCOMES:
Implantation rate | 4 weeks
  The ratio of embryo implantation measured through ultrasound
Pregnancy rate | 6 weeks
  The ratio of pregnancy measured through βHCG

CONTACTS AND LOCATIONS:
Overall Officials: Nikica Zaninovic, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Center for Reproductive Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No